CLINICAL TRIAL: NCT05521672
Title: Clinical Trial Phase IIa to Evaluate the Safety and Effectiveness of Treatment With Fat-derived Mesenchymal Allogenic Mesenchymal Troncal Cells in Patients With Single Inflammatory Stenosis in the Context of Crohn's Disease.
Brief Title: Clinical Trial to Evaluate if the Laparoscopic Administration of Cells Derived From the Fatty Tissue Can Improve the Inflammatory Stenosis in Patient With Crohn's Disease
Acronym: MEIC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: low recruitment
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Effice Servicios Para la Investigacion S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FJD-MEIC-21-01; 2021-006068-26 (EudraCT Number)
Record Dates: First submitted 2022-08-22; First posted 2022-08-30 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Stenosis; Bowel; Crohn Disease
MeSH Terms: conditions — Constriction, Pathologic; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Dose (Experimental): This is an uncontrolled trial, phase IIa, proof of concept. Group control has not been included.
  All patients will receive one single dose of 120 million cells
  Interventions: Drug: Adipose derived allogenic mesenchymal stem cells (adAMSC)

INTERVENTIONS:
Drug: Adipose derived allogenic mesenchymal stem cells (adAMSC) — adAMSC will be administered in the perilesional adipose tissue, through a laparoscopic procedure

SUMMARY:
A phase II, national, multicenter, uncontrolled and open trial to evaluate the feasibility and safety of laparoscopic administration of adipose derived allogenic mesenchymals stem cells (adMSC), for the treatment of patients with a single inflammatory stenosis in the context of Crohn's disease.

DETAILED DESCRIPTION:
The hypothesis of the study is that the drug study administration will result in a anti-inflammatory effect, preventing the progression of the stenotic lesion and thus reducing the need to perform surgical resections.

A multicentre, national, uncontrolled and open-label pilot study will be performed. 20 adult patients fulfilling eligibility criteria will be included.

The trial is organized in screening period, treatment period and 6 follow-up visits.

The treatment visit will be done in operating theatre, as the study drug is administrated by laparoscopy with a total dose of 120 million cells prepared in a saline solution with a cell concentration of 10 million cells per millilitre.

Follow-up visits are divided into 4 visits that will take place every 6 weeks (+-7 days) until week 24; 1 additional follow-up visit will take place at week 36 and the last one at week 52.

Analytical controls (blood count, biochemistry and coagulation) will be carried out throughout the trial and biological samples will be taken in three visits (Screening, visit 3 and visit 6).

Abdominal MRI will be performed at baseline and in the end of study visit, to assess stenosis evolution.

The overall duration of the trial is 36 months from the start of recruitment to the last follow-up visit. The period planned for this trial is from september 2022 to september 2025.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who agree to participate and agree to give their written consent.
2. Patients older than 18 years and younger than 75 years
3. With Crohn's disease diagnosed at least 6 months before that meet clinical, endoscopic, histological and/or radiological criteria.
4. Presence of a single inflammatory stenotic lesion in the small intestine or ileocolic area with a maximum length of 5 cm, demonstrated by magnetic resonance enterography, which produces episodes of intestinal occlusion/subocclusion. Other inflammatory lesions are admittedly present, but only one should be identified as the obvious cause of the occlusion/subocclusion.
5. Patients treated with at least one biological drug and with inadequate response to maintenance doses and before intensification (either dose, interval or change/addition of another drug):

   1. antiTNF (for at least 14 week, include induction and/or maintenance doses): Infliximab, Adalimumab, Certolizumab.
   2. Anti-integrin (for at least 14 week, include induction and/or maintenance doses): Vedolizumab
   3. Anti-IL-12/23 (for at least 16 week, include induction and/or maintenance doses): Ustekinumab
6. Women of childbearing potential must have a negative pregnancy test at screening and agree to use effective contraceptive measures for the duration of their participation in the study*

   * a woman is considered to be of childbearing potential (WOCBP), that is, fertile, after menarche and until she becomes postmenopausal, unless she is permanently infertile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.

Highly effective methods are considered: combined hormonal contraception (containing estrogens and progestogens) associated with ovulation inhibition (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with ovulation inhibition (oral, injectable, implantable ), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner, sexual abstinence

Exclusion Criteria:

1. Intra-abdominal abscesses larger than 3 cm not drained (surgically, by interventional radiology) or not treated with antibiotics. Patients may be included once the abscess has been drained (without the need to wait) or if they have received antibiotic treatment, once improvement has been confirmed with imaging tests.
2. Several intestinal obstruction that requires urgent surgery
3. Active outbreak of Crohn's disease requiring medical treatment, defined as abdominal pain, fever, bloody diarrhea and CRP greater than 10. The patient may be included once the condition has resolved, when the patient is on maintenance medication.
4. History of previous invasive neoplasia in the last 5 years. Patients with completely resected basal cell carcinoma of the skin may be included
5. History in the last 6 month of several, progressive or uncontrolled hepatic, hematological, gastrointestinal, renal, endocrine, pulmonary, cardiac, neurological or psychiatric disease
6. Patients with primary sclerosing cholangitis
7. Patients with known congenital or acquired immunodeficiency, including HIV
8. Known allergy or hypersensibility to penicillin or aminoglycosides; DMEN (dulbecco modified eagle´s medium), bovine serum, local anesthesic or gadolinium
9. Contraindication to perform MRI (pacemaker, hip replacement or severe claustrophobia).
10. Patients unwilling or unable to comply with study procedures.
11. Patients who are receiving or have received any investigational drug in the 3 months prior to the screening period
12. Major surgery or severe trauma in the previous 6 months.
13. Pregnant or lactating women.
14. Patients who have a contraindication for general anesthesia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Percentage of complications | Through study completion, an average of 2 years
  Number of complication associated with presurgery, surgery, IMP administration and postsurgery period
Change from baseline length and diameter of the stenosis | From screening visit to week 52
  according to RMI
Crohn's disease activity index (CDAI) questionnaire score | Through study completion, an average of 2 years
  Change from baseline in Crohn's disease activity index (CDAI) score (0-1100 points).
  Higher scores mean a worse outcome.
inflammatory bowel disease questionnaire (IBDQ32 ) | Through study completion, an average of 2 years
  Change from baseline in inflammatory bowel disease questionnaire (IBDQ32 ). 140-200 points, higher scores mean a better outcome.
patients with an obstructive episode who required resection surgery | Through study completion, an average of 2 years
  number of patients with an obstructive episode who required resection surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Herreros, Principal Investigator — Hospital Fundación Jiménez Diaz
Locations (3):
- Spain (3):
  - Hospital Universitario Valle de Hebrón, Barcelona
  - Hospital Universitario Fundación Jiménez Diaz, Madrid
  - Hospital Universitario y Politécnico La Fe, Valencia